CLINICAL TRIAL: NCT05259670
Title: Risk Factors for Recurrent Intussusception After Successful Reduction in Pediatric Patients in a Tertiary Care Hospital of Nepal: A Prospective-Study
Brief Title: Risk Factors for Recurrent Intussusception Successful Reduction in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Sanjeev Kharel (Other)
Collaborators: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Sponsor-Investigator, Sanjeev Kharel, Sponsor investigator, Nepal Medical Student Society
Organization: Nepal Medical Student Society (Other)
Other Study IDs: 077/078
Record Dates: First submitted 2022-02-16; First posted 2022-02-28 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Intussusception
Keywords: Hydrostatic reduction; Recurrence; Pediatrics
MeSH Terms: conditions — Intussusception; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine risk factors associated with recurrent intussusception among pediatric patients who have undergone successful reduction at a tertiary care hospital.

DETAILED DESCRIPTION:
This is the prospective observational study. In this study, 78 patients,age <16 years with diagnosis of intussusception between June 2019 and April 2020 who had successful reduction with either hydrostatic reduction and/or operative reduction in Teaching Hospital were enrolled in the study. They were followed up to a period of 1 month for recurrence of intussusception. The recurrent cases were thus identified and various variables were compared between recurrent and non-recurrent cases by univariable and multivariable analysis.

This prospective observational study was approved by the ethics committees of Institutional review board of Tribhuvan University, Institute of Medicine.

A standard structured questionnaire was filled by interviewing the patient (if possible) and family members/relatives after taking informed written consent. The questionnaire documented the patient's age, sex, weight, duration of symptoms, presenting symptoms: abdominal pain, excessive cry, vomiting, lethargy, blood in stool, fever, palpable mass, constipation, diarrhoea ,location of mass, enlarged lymph nodes(LNs), blood counts and methods of reduction. Age of 2 years, weight of 12 kg and duration of symptoms of 48 hours was used to classify patients into two groups

ELIGIBILITY:
Inclusion Criteria:

* We included the patients who were diagnosed with intussusception from the age of 0 year to 16 years who received nonoperative and operative reduction as an initial treatment.

Exclusion Criteria:

* Pediatric patients with spontaneous reduction of hydro-reduction and who required resection and anastomosis as a part of operative procedure were excluded from the study.

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric population age less than 16 years old recruited undergoing recurrent intussusception with successful reduction followed up for 1 month.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Risk factor for recurrent intussusception | June 2019-April 2020
  Significant risk factor for recurrent intussusception after successful reduction

CONTACTS AND LOCATIONS:
Locations (2):
- Nepal (2):
  - Tribhuvan University Teaching hospital, Kathmandu, Bagmati
  - Tribhuvan University Teaching hospital, Maharajgunj, Bagmati